CLINICAL TRIAL: NCT05659810
Title: The Effect of Preoperative Gabapentin on the Duration of Spinal Anesthesia in Patients Undergoing Lower Limb Surgery: A Double-blind, Randomized Clinical Study
Brief Title: The Effect of Gabapentin on Spinal Anesthesia Duration
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Refaat, Lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R 177/2022
Record Dates: First submitted 2022-11-23; First posted 2022-12-21 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Prolongation of Spinal Anesthesia
Keywords: Gabapentin, Spinal, Anesthesia, Visual analogue scale
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Randomization by concealed envelope method
Who Masked: Participant, Outcomes Assessor
Masking Description: A physician assessing outcomes blinded to the nature of the study and will monitor the block density and regression time. Drugs will be given to the patient by an anesthesiologist unaware of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative oral gabapentin before spinal anesthesia (Active Comparator): The participants will receive 900 mg of gabapentin before surgery in 2 divided doses; 300 mg 10 hours prior to surgery and 600 mg 2 hours before surgery.
  Interventions: Drug: Gabapentin 300mg
- Preoperative oral placebo before spinal anesthesia (Placebo Comparator): The participants will receive 1 tablet 10 hours prior to surgery, and then 2 tablets 2 hours prior to surgery
  Interventions: Drug: Gabapentin 300mg

INTERVENTIONS:
Drug: Gabapentin 300mg — Preoperative gabapentin before spinal anesthesia
  Other Names: placebo tablet

SUMMARY:
This prospective parallel group double blinded randomized study will be conducted over 60 adult participants between 20 and 60 years ASA (American Association of Anesthesiologists) I and II. The participants will be randomly allocated in 2 groups. Group A will receive 900 mg of gabapentin before surgery in 2 divided doses; 300 mg 10 hours prior to surgery and 600 mg 2 hours before surgery, while group B will receive 2 placebo tablets at the same time. The participants will receive spinal anesthesia in the form of 3ml of hyperbaric bupivacaine 0.5%. Hemodynamics will be recorded every 15 minutes till the end of surgery. Sensory, and motor block progression, and regression will be recorded also.

DETAILED DESCRIPTION:
A prospective double blinded randomized trial to study the effect of gabapentin on the duration of spinal anesthesia. The participants will be divided into 2 groups. Group A will receive 900 mg of gabapentin before surgery in 2 divided doses; 300 mg 10 hours prior to surgery and 600 mg 2 hours before surgery, while group B will receive 2 placebo tablets at the same time.

The patient will be seated and after sterilization of his back with povidone iodine, a midline intrathecal injection of the 3ml of hyperbaric bupivacaine 0.5% at L 3/4 - L4/5 will be done via a 25G needle. Neural block will be assessed by using pin prick test, motor block will be assessed by using the modified Bromage scale, results will be recorded every 3 min until the level is stable for 3 consecutive tests.

After successful intrathecal injection, the patient will be monitored continuously for block progression and complications. The patient's blood pressure will be taken every 3 minutes initially, more frequently if needed. The patient will be monitored for the following:

Ensure that the block is adequate for the surgical procedure and it does not progress too high (motor block will be assessed by modified Bromage score and the sensory level by pin prick test up to T7-T10 level)

Sensory block will be assessed by pin prick test (Hollman test) using a 3-point scale; (0) = Normal sensation, (1) = Loss of sensation of pin prick (analgesia), and (2) = Loss of sensation of touch (anesthesia).

Onset time for sensory block will be defined as the time interval between the end of local anesthetic administration and complete sensory block (score 2 for all nerves). Duration of sensory block will be defined as the time interval between the complete sensory block and complete resolution of anesthesia (score 0 for all nerves).

Motor block is determined by using the modified Bromage scale (Bromage 0, the patient is able to move the hip, knee and ankle; Bromage 1 when the patient is unable to move the hip but is able to move the knee and ankle, Bromage 2 when the patient is unable to move the hip and knee but able to move the ankle, Bromage 3 when the patient is unable to move the hip, knee and ankle). The interval between the injection and block completion was considered as the onset of motor block. Duration of motor block will be defined as the time interval between the complete motor block and complete resolution of anesthesia. Failed block will be considered if the sensory block and motor block were not achieved after 20 min.

- Pain assessment: Patients will be followed every 2 hours postoperatively till 12 hours for analgesic requirements. Postoperative pain will be assessed via the Visual analogue scale (VAS), and when the VAS is more than 4 the patient will receive 0.25mg/kg nalbuphine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I, and II
* Age 20 - 60 years
* Weight between 60 and 80 kilograms
* Height between 160 and 180 centimetres

Exclusion Criteria:

* Participants with contraindications to spinal anesthesia.
* Participant refusal
* Extreme short or tall statures
* Body mass index above 40

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the time of regression of sensory block | 4 hours
  Measurement of the time of regression of sensory block by using pin prick test
Measurement of time of regression of motor block | 4 hours
  Measurement of time of regression of motor block by using Bromage scale from 0-4

SECONDARY OUTCOMES:
Measurement of time to onset of sensory block | 15 minutes
  Measurement of time to onset of sensory block by using pin prick test
Measurement of duration of postoperative analgesia | 12 hours
  Measurement of the duration of postoperative analgesia using the visual analogue scale from 0-10

OTHER OUTCOMES:
Amount of postoperative analgesics required | 24 hours
  Measurement of the number of doses needed of postoperative analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Ain Shams, Principal Investigator — University Hospital
Locations (1):
- Ain Shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No